CLINICAL TRIAL: NCT02995733
Title: Patient Empowered Strategy to Reduce Asthma Morbidity in Highly Impacted Populations
Brief Title: Patient Empowered Strategy to Reduce Asthma Morbidity in Highly Impacted Populations; PeRson EmPowered Asthma RElief
Acronym: PREPARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); American Academy of Family Physicians (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016P001839
Record Dates: First submitted 2016-11-09; First posted 2016-12-16 (Estimated); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Asthma
Keywords: asthma; African Americans; Hispanics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PARTICS (Active Comparator): addition of PARTICS strategy - Patient Activated Reliever-Triggered Inhaled CorticoSteroid (PARTICS) using QVAR . Patient will use inhaled corticosteroid at time of rescue inhaler use
  Interventions: Drug: PARTICS using QVAR
- Usual Care (No Intervention): Provider-enhanced usual care arm; no change in asthma management

INTERVENTIONS:
Drug: PARTICS using QVAR — Patient takes inhaled corticosteroid at the time of rescue inhaler use
  Other Names: Patient Activated Reliever-Triggered Inhaled CorticoSteroid
  Arms: PARTICS

SUMMARY:
Asthma imposes a significant burden in the US in terms of morbidity, costs to society, individual suffering, loss of productivity and mortality. African Americans (AA) and Hispanic/Latinos (H/L) bear a disproportionate share of that morbidity. Despite national guidelines for asthma treatment, the gap between these groups and whites has been stable or widening. The need for pragmatic research to address the continuing burden is widely recognized. Patients use asthma reliever inhalers to provide immediate relief of symptoms. Controller inhalers (inhaled corticosteroids (ICS)) are intended to be used regularly to prevent symptoms and attacks. Guidelines suggest that they be used daily, on a fixed basis, in all but the mildest asthma. However, adherence by patients and implementation of evidence-based guideline recommendations by clinicians has been poor. Gap analysis suggests that it is difficult to improve adherence to the current recommendations without complex and resource-intensive interventions. Studies have examined symptom-activated use of ICS triggered by use of a reliever medication. The Investigators call this approach PARTICS - Patient Activated Reliever-Triggered Inhaled CorticoSteroid. Explanatory, non-real world studies suggest that PARTICS can produce up to 50% reductions in asthma attacks compared with usual care, while reducing ICS use by half or more. These studies have been performed in pre-selected populations, which represent less than 5% of asthma patients. The previous studies have been done with repeated education and adherence checks in both the intervention and control arms.

The investigators have consulted with AA and H/L patients, health care providers, leaders of professional societies, advocacy groups, health policy leaders, pharmacists, and pharmaceutical manufacturers. All groups have indicated that asthma decision making would be changed if we demonstrated that implementing PARTICS improves important asthma outcomes such as reducing exacerbations. The Investigators have designed a study with the stakeholders to determine whether PARTICS can improve outcomes that are important to patients when superimposed on a background provider-educated standard of care through the Asthma IQ system. The Investigators propose a study entitled PREPARE: Patient Empowered Strategy to Reduce Asthma Morbidity in Highly Impacted Populations. The Investigators aim to determine whether PARTICS can reduce asthma morbidity in AA and H/L.

DETAILED DESCRIPTION:
Asthma imposes a significant burden on the US population in terms of morbidity, costs to society, individual suffering, loss of productivity and mortality. African Americans (AA) and Hispanic/Latinos (H/L) bear a disproportionate share of that morbidity. Despite introduction of national guidelines for asthma treatment, the gap between these groups and whites has been stable or widening. The need for pragmatic research to address the continuing burden is widely recognized. Patients use asthma reliever inhalers to provide immediate relief of symptoms. Controller inhalers (inhaled corticosteroids (ICS)) are intended to be used regularly to prevent symptoms and attacks. Guidelines suggest that they be used daily, on a fixed basis, in all but the mildest asthma. However, adherence by patients and implementation of evidence-based guideline recommendations by clinicians has been poor. Gap analysis suggests that it is difficult to improve adherence to the current recommendations without complex and resource-intensive interventions.

Studies have examined symptom-activated use of ICS triggered by use of a reliever medication. We call this approach PARTICS - Patient Activated Reliever-Triggered Inhaled CorticoSteroid. Explanatory, non-real world studies suggest that PARTICS can produce up to 50% reductions in asthma attacks compared with usual care, while reducing ICS use by half or more. However, these studies have been performed in pre- selected populations, which represent less than 5% of patients with asthma. They have been done with repeated education and adherence checks in both the intervention and control arms.

The investigators have consulted with AA and H/L patients, health care providers, leaders of professional societies, advocacy groups, health policy leaders, pharmacists, and pharmaceutical manufacturers. All groups have indicated that asthma decision making would be changed if it was demonstrated that implementing PARTICS improves important asthma outcomes such as reducing rates of exacerbations. Together with our partners and stakeholders, the investigators have designed a study to determine whether PARTICS can improve outcomes that are important to patients when superimposed on a background provider-educated standard care through the Asthma IQ system. The investigators therefore propose a study entitled PREPARE: Patient Empowered Strategy to Reduce Asthma Morbidity in Highly Impacted Populations. The aim is to determine whether a PARTICS strategy can reduce asthma morbidity in AA and H/L. The primary outcome will be asthma exacerbations which have been shown to be important to patient and healthcare stakeholders. The secondary outcomes will include additional outcomes important to patients (i.e. days lost from work or school, asthma control, & asthma quality of life). The investigators have broad input and involvement from multiple stakeholder groups in study design, implementation, and commitments for dissemination. AA and H/L patients and their advocates have been involved and will continue to play a central role in all phases of the study.

ELIGIBILITY:
INCLUSION CRITERIA

* Black or Hispanic based on self-identification (Hispanic if identify as both)
* Male and female, ages 18-75 years
* Ability to provide informed consent
* Clinical history consistent with asthma for > 1 year.
* Prescribed ICS as daily maintenance therapy
* Participant must also have an ACT score of 19 or less, or a history of one or more exacerbations in the past year that required patient report of systemic corticosteroid use.

EXCLUSION CRITERIA

* Life expectancy less than one year
* Known allergy to the ICS inhaler used in the study
* Having COPD or other chronic lung disease other than asthma; with the exception of the following:

  * Dx of COPD in a never smoker without any other lung disease or any other disease that might cause airway obstruction such as: Cystic Fibrosis, Connective Tissue Disease, premature birth, organ transplantation, bronchiectasis, sarcoid, and obliterative bronchiolitis
  * Dx of COPD in former smoker with normal PFTs done after the person quit smoking
  * Dx of COPD in current smoker with normal PFTs done in past 24 months
  * Dx of COPD IN CURRENT OR FORMER SMOKER with obstruction on PFTs: normal diffusing capacity in past 24 months and demonstrated reversibility of 12% or more at any time
* Regular systemic corticosteroid use daily or every other day for any reason-including asthma or other medical reasons
* Use of systemic corticosteroid, or visit to the doctor's office, emergency department (ED) or urgent care, or overnight hospitalization for an asthma exacerbation in the past month (can wait and re-check eligibility after one month)
* Use of biologics (injections or infusion medicines): with the exception of the following:

  * the patient has been on a stable dose of a biologic for at least 6 months and,
  * must have had an exacerbation at least 2 months after starting on a biologic to be considered eligible OR
  * must have a current ACT score <=19 to be considered eligible.
* Bronchial thermoplasty less than 6 months ago (can re-check eligibility 6 months after procedure)
* Another family member living in the same household already enrolled in study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (20):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Grace Medical Home, Orlando, Florida
  - University of Central Florida, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - University of Illinois- Chicago, Chicago, Illinois
  - Baystate Health Center, Springfield, Massachusetts
  - Mt. Sinai, New York, New York
  - Montefiore, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - MetroHealth, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Callen E, Israel E, Cardet JC, Fuhlbrigge AL, Manning B, Gaona G, Staton E, Pace WD. Electronic health record data analysis on the impact of rescue-triggered inhaled corticosteroids on controller therapy in Black and Latinx individuals from a pragmatic, open-label, patient-level randomised trial. BMJ Open. 2024 Nov 21;14(11):e088349. doi: 10.1136/bmjopen-2024-088349. PMID 39578039
- [Derived] Ishmael L, Apter A, Busse PJ, Calderon-Candelario R, Carroll JK, Casale T, Celedon JC, Cohen R, Coyne-Beasley T, Cui J, Ericson B, Hernandez P, Kaelber DC, Maher N, Merriman C, Mosnaim G, Nazario S, Phipatanakul W, Pinto-Plata V, Riley I, Shenoy K, Wisnivesky J, Yawn B, Israel E, Cardet JC. Asthma morbidity measures across Black ethnic subgroups. J Allergy Clin Immunol. 2024 Feb;153(2):408-417. doi: 10.1016/j.jaci.2023.10.028. Epub 2023 Nov 23. PMID 38000696
- [Derived] Ugalde IC, Ratigan A, Merriman C, Cui J, Ericson B, Busse P, Carroll JK, Casale T, Celedon JC, Coyne-Beasley T, Fagan M, Fuhlbrigge AL, Villarreal GG, Hernandez PA, Jariwala S, Kruse J, Maher NE, Manning B, Mosnaim G, Nazario S, Pace WD, Phipatanakul W, Pinto-Plata V, Riley I, Rodriguez-Louis J, Salciccioli J, Shenoy K, Shields JB, Tarabichi Y, Sosa BT, Wechsler ME, Wisnivesky J, Yawn B, Israel E, Cardet JC. Preference for and impact of telehealth vs in-person asthma visits among Black and Latinx adults. Ann Allergy Asthma Immunol. 2023 Nov;131(5):614-627.e2. doi: 10.1016/j.anai.2023.07.012. Epub 2023 Jul 23. PMID 37490981
- [Derived] Forth VE, Cardet JC, Chang KL, Ericson B, Hurley LP, Maher NE, Staton EW, Sosa BT, Israel E; PREPARE investigators. What Patients Call Their Inhalers Is Associated with "Asthma Attacks". J Am Board Fam Med. 2023 Aug 9;36(4):650-661. doi: 10.3122/jabfm.2022.220270R2. Epub 2023 Jul 19. PMID 37468217
- [Derived] Cardet JC, Shenoy K, Baydur A, Carroll JK, Celedon JC, Cui J, Dara P, Ericson B, Forth VE, Fagan M, Fuhlbrigge AL, Gupta R, Hart MK, Hernandez ML, Hernandez PA, Kruse J, Maher NE, Manning BK, Pinto-Plata VM, Robles J, Rodriguez-Louis J, Shields JB, Telon Sosa BS, Wechsler ME, Israel E. Caribbean Latinx with moderate-severe asthma bear greater asthma morbidity than other Latinx. J Allergy Clin Immunol. 2022 Nov;150(5):1106-1113.e10. doi: 10.1016/j.jaci.2022.05.026. Epub 2022 Jun 30. PMID 35779669
- [Derived] Israel E, Cardet JC, Carroll JK, Fuhlbrigge AL, She L, Rockhold FW, Maher NE, Fagan M, Forth VE, Yawn BP, Arias Hernandez P, Kruse JM, Manning BK, Rodriguez-Louis J, Shields JB, Ericson B, Colon-Moya AD, Madison S, Coyne-Beasley T, Hammer GM, Kaplan BM, Rand CS, Robles J, Thompson O, Wechsler ME, Wisnivesky JP, McKee MD, Jariwala SP, Jerschow E, Busse PJ, Kaelber DC, Nazario S, Hernandez ML, Apter AJ, Chang KL, Pinto-Plata V, Stranges PM, Hurley LP, Trevor J, Casale TB, Chupp G, Riley IL, Shenoy K, Pasarica M, Calderon-Candelario RA, Tapp H, Baydur A, Pace WD. Reliever-Triggered Inhaled Glucocorticoid in Black and Latinx Adults with Asthma. N Engl J Med. 2022 Apr 21;386(16):1505-1518. doi: 10.1056/NEJMoa2118813. Epub 2022 Feb 26. PMID 35213105
- [Derived] Cardet JC, Busse PJ, Carroll JK, Casale TB, Coyne-Beasley T, Dixon-Williams S, Fagan M, Forth VE, Fuhlbrigge AL, Hernandez ML, Kaelber D, Kaplan B, Lorenzi M, Madison S, Maher NE, Majewski K, Manning B, McKee MD, Nazario S, Pace WD, Pencina MJ, Rand CS, Rodriguez-Louis J, She L, Shields J, Teng JE, Wechsler ME, Wisnivesky JP, Yawn BP, Israel E. Adherence to adding inhaled corticosteroids to rescue therapy in a pragmatic trial with adults with asthma: A pilot study. Ann Allergy Asthma Immunol. 2020 May;124(5):487-493.e1. doi: 10.1016/j.anai.2019.12.027. Epub 2020 Jan 8. PMID 31923550

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1220 participants were enrolled, however, 19 participants were not followed and were dropped from analysis due to the site closure. They were not included in the primary analyses but were included in safety reporting. Two sites were enrolling simultaneously and there was one additional participant enrolled accidentally.
Period: Overall Study
Arm/Group | PARTICS | Usual Care
Started | 609 | 611
Completed | 542 | 557
Not Completed | 67 | 54
Not completed — Study site closed | 9 | 10
Not completed — Death | 3 | 4
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Removed by study team due to inappropriate behavior | 1 | 0
Not completed — Lost to Follow-up | 48 | 37
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: 19 participants were dropped from analysis due to the site closure. They were not followed and not included in any analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | PARTICS | Usual Care | Total
Number analyzed (Participants) | 600 | 601 | 1201
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.5) | 47.0 (13.9) | 47.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 508 | 497 | 1005
  Male | 92 | 104 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: African American/Black | 303 | 300 | 603
  Race/ethnicity: Hispanic/Latinx | 297 | 301 | 598
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 51 | 51 | 102
  United States | 549 | 550 | 1099
Body mass index (BMI) (kg/m2) [Mean (Standard Deviation); unit: kilograms per meters squared] | 35.2 (9.1) | 35.1 (9.5) | 35.1 (9.3)
Obesity [Count of Participants; unit: Participants] — The body-mass index is the weight in kilograms divided by the square of the height in meters. Obesity was defined as a body-mass index of 30 or higher.
  Participants | 421 | 403 | 824
Smoking status [Count of Participants; unit: Participants] — Current smokers were defined as participants who were currently smoking or had smoked within the previous year. Former smokers were participants who had not smoked in the previous year but had smoked at least 10 pack-years. Nonsmokers were those who had not smoked within the previous year and had smoked less than 10 pack-years.
  Participants
    Current smoker | 69 | 74 | 143
    Former smoker | 54 | 46 | 100
    Non-smoker | 477 | 481 | 958
Nonsmoker or former smoker in smoking environment [Count of Participants; unit: Participants] — A smoking environment was defined as others regularly smoking in the participant's home, work, or car.
  Participants | 96 | 107 | 203
Number of pack-years of smoking [Mean (Standard Deviation); unit: pack-years] — Population: 376 participants answered questions about smoking pack-years. Non-smokers are those who have not smoked within 1 year and have smoked less than 10 pack-years in their lifetime. 143 are current smokers, 100 are former smokers, and 133 are non-smokers with less than 10 pack-years.
  pack-years
    number analyzed (Participants) | 190 | 186 | 376
    (all) | 12.4 (13.80) | 15.8 (19.79) | 14.1 (17.09)
Maintenance asthma medications: Inhaled glucocorticoid without long-acting beta-agonist [Count of Participants; unit: Participants] — Medication categories are not mutually exclusive and therefore are reported separately.
  Participants | 171 | 169 | 340
Maintenance asthma medications: Combination inhaled glucocorticoid with long-acting beta-agonist [Count of Participants; unit: Participants] — Medication categories are not mutually exclusive and therefore are reported separately.
  Participants | 428 | 431 | 859
Maintenance asthma medications: Long-acting muscarinic antagonist [Count of Participants; unit: Participants] — Medication categories are not mutually exclusive and therefore are reported separately.
  Participants | 64 | 79 | 143
Maintenance asthma medications: Leukotriene-receptor antagonist [Count of Participants; unit: Participants] — Medication categories are not mutually exclusive and therefore are reported separately.
  Participants | 308 | 290 | 598
Maintenance asthma medications: Biologic agent [Count of Participants; unit: Participants] — Medication categories are not mutually exclusive and therefore are reported separately. Biologic agents included injectable monoclonal antibody therapies targeting IgE, interleukin-5 or the interleukin-5 receptor, or the interleukin-4 receptor.
  Participants | 17 | 19 | 36
Use of quick-reliever nebulizer [Count of Participants; unit: Participants] | 408 | 396 | 804
Number of quick-reliever nebulizations per week [Mean (Standard Deviation); unit: Nebulizations per week] — Population: Only participants who reported using a nebulizer are included in this measure.
  Nebulizations per week
    number analyzed (Participants) | 408 | 396 | 804
    (all) | 2.7 (4.6) | 3.0 (4.8) | 2.9 (4.7)
Number of coexisting conditions [Count of Participants; unit: Participants] — Coexisting conditions included heart disease, cancer (except skin cancer), stroke, diabetes, chronic kidney disease, chronic obstructive pulmonary disease, human immunodeficiency virus infection or acquired immunodeficiency syndrome, hypertension, depression, and sleep disorder.
  Participants
    0 | 166 | 191 | 357
    1 | 150 | 126 | 276
    2 | 133 | 119 | 252
    3 | 81 | 86 | 167
    4 or more | 70 | 79 | 149
Fractional exhaled nitric oxide (FeNO) [Mean (Standard Deviation); unit: ppb] — Population: 1003 participants had FeNO data available for analysis.
  ppb
    number analyzed (Participants) | 502 | 501 | 1003
    (all) | 26.7 (27.8) | 30.4 (34.9) | 28.6 (31.6)
Fractional exhaled nitric oxide (FeNO), ≥30 ppb [Count of Participants; unit: Participants] — Population: 1003 participants had FeNO data available for analysis.
  Participants
    number analyzed (Participants) | 502 | 501 | 1003
    (all) | 148 | 154 | 302
Absolute eosinophil count [Mean (Standard Deviation); unit: cells/μL] — Population: 996 participants had eosinophil count data available for analysis.
  cells/μL
    number analyzed (Participants) | 502 | 494 | 996
    (all) | 245.5 (229.29) | 250.1 (247.48) | 247.8 (238.47)
Absolute eosinophil count [Median (Full Range); unit: cells/μL] — Population: 996 participants had eosinophil count data available for analysis.
  cells/μL
    number analyzed (Participants) | 502 | 494 | 996
    (all) | 188 [0 to 1938.8] | 195 [0 to 3555.9] | 192 [0 to 3555.9]
Absolute eosinophil count ≥300 cells/μL [Count of Participants; unit: Participants] — Population: 996 participants had eosinophil count data available for analysis.
  Participants
    number analyzed (Participants) | 502 | 494 | 996
    (all) | 128 | 137 | 265
History of ≥1 asthma exacerbation in past year [Count of Participants; unit: Participants] — Asthma exacerbation in the previous year was defined as a participant-reported emergency department or urgent care visit, hospitalization, or course of systemic glucocorticoids within the 12 months before randomization.
  Participants | 440 | 427 | 867
Asthma Control Test score [Mean (Standard Deviation); unit: units on a scale] — The Asthma Control Test is a participant-administered tool for assessing the level of asthma control.Total scores range from 5 to 25, with a score of 20 to 25 indicating well-controlled asthma, a score of 16 to 19 indicating asthma that was not well controlled, and a score of 5 to 15 indicating very poorly controlled asthma. The minimal clinically important difference is 3 points.
  units on a scale | 14.7 (4.4) | 14.5 (4.5) | 14.6 (4.4)
Asthma Symptom Utility Index score [Mean (Standard Deviation); unit: units on a scale] — The Asthma Symptom Utility Index is a participant-administered tool for assessing preference-based quality of life. Scores range from 0 (worst possible symptoms) to 1 (no symptoms). The minimal clinically important difference is 0.09. Population: One participant in the Usual Care group is missing baseline ASUI data.
  units on a scale
    number analyzed (Participants) | 600 | 600 | 1200
    (all) | 0.67 (0.22) | 0.67 (0.21) | 0.67 (0.21)
Medication Adherence Report Scale-5 score [Mean (Standard Deviation); unit: units on a scale] — The Medication Adherence Report Scale-5 measures participant-reported medication adherence. Mean scores are calculated from five items and range from 1 to 5, with higher scores indicating better adherence.
  units on a scale | 4.2 (0.8) | 4.2 (0.8) | 4.2 (0.8)
Low or marginal health literacy [Count of Participants; unit: Participants] — Health literacy was assessed with the Brief Health Literacy Scale, which measures participant-reported health literacy and consists of three items. Scoring low or marginal health literacy on any one item classifies a participant as having low or marginal health literacy. Population: One participant in the PARTICS group is missing baseline data measuring health literacy.
  Participants
    number analyzed (Participants) | 599 | 601 | 1200
    (all) | 101 | 100 | 201
Participant-perceived overall health [Count of Participants; unit: Participants]
  Excellent | 13 | 9 | 22
  Very good | 68 | 60 | 128
  Good | 200 | 194 | 394
  Fair | 257 | 272 | 529
  Poor | 62 | 66 | 128

OUTCOME MEASURES:

1. Primary Outcome: Rate of Asthma Exacerbations Per Year
Description: Our primary outcome, the rate of asthma exacerbations per year, is defined as the number of exacerbations, emergency room visits, or hospitalizations requiring oral or parenteral corticosteroids, per patient per year
Time Frame: monthly through study completion an average of 15 months
Measure: Mean (95% Confidence Interval); unit: Adjusted annualized exacerbations
Arm/Group | PARTICS | Usual Care
Number analyzed (Participants) | 600 | 601
Adjusted annualized exacerbations | 0.69 [0.61 to 0.78] | 0.82 [0.73 to 0.92]
Statistical Analysis 1: Comparison: PARTICS vs Usual Care; Test type: Superiority — Asthma exacerbation rates during follow-up between two randomized treatment arms are compared using the Andersen-Gill adaptation of time-to-event Cox proportional hazard model with robust standard errors to account for multiple occurrences of the outcome in each patient (Andersen Gill, 1982). This analysis is based on intention-to-treat (ITT) patient population; p = 0.048, Cox proportional hazard model; Pre-specified baseline covariates are adjusted in the model. A time-dependent covariate for the COVID pandemic is also included in adjustments; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.720 to 0.999]

2. Secondary Outcome: Asthma Control: Asthma Control Test (ACT) Score, Least-squares Mean Change From Baseline
Description: Asthma control represents the degree to which impairment (impact of asthma on patient's daily life) is minimized and the goals of therapy are met. The Asthma Control Test is a participant-administered tool for assessing the level of asthma control. Total scores range from 5 to 25, with a score of 20 to 25 indicating well-controlled asthma, a score of 16 to 19 indicating asthma that was not well controlled, and a score of 5 to 15 indicating very poorly controlled asthma. The minimal clinically important difference is 3 points
Time Frame: Monthly through study completion an average of 15 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PARTICS | Usual Care
Number analyzed (Participants) | 600 | 601
units on a scale | 3.4 [3.1 to 3.6] | 2.5 [2.3 to 2.8]
Statistical Analysis 1: Comparison: PARTICS vs Usual Care; Test type: Superiority — Mixed model is used to compare the treatment effects. The response variable is ACT change at each monthly assessment from baseline. The covariates (included as fixed effects) include randomized treatment arm, continuous time of assessment as a linear and quadratic term and the interactions of the treatment arm with the time variables. Independent random effects include intercept and time variables. The model adjusts for all the baseline covariates included in the primary analysis; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.5 to 1.2]

3. Secondary Outcome: Preference Based Quality of Life: Asthma Symptom Utility Index (ASUI), Least-squares Mean Change From Baseline
Description: The ideal outcome measure for any comparative effectiveness analysis captures the risks and benefits for each of the interventions from the patient's point of view. The use of a preference-based instrument, the Asthma Symptom Utility Index (ASUI), captures this important information. The Asthma Symptom Utility Index is a participant-administered tool for assessing preference-based quality of life. Scores range from 0 (worst possible symptoms) to 1 (no symptoms). The minimal clinically important difference is 0.09.
Time Frame: Monthly through study completion an average of 15 months
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PARTICS | Usual Care
Number analyzed (Participants) | 600 | 601
units on a scale | 0.12 [0.11 to 0.13] | 0.08 [0.07 to 0.09]
Statistical Analysis 1: Comparison: PARTICS vs Usual Care; Test type: Superiority — Mixed model is used to compare the treatment effects. The response variable is ASUI change at each monthly assessment from baseline. The covariates (included as fixed effects) include randomized treatment arm, continuous time of assessment as a linear and quadratic term and the interactions of the treatment arm with the time variables. Independent random effects include intercept and time variables. The model adjusts for all the baseline covariates included in the primary analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [0.02 to 0.05]

4. Secondary Outcome: Days Per Year Lost From Work or School/ Days Unable to Carry Out Usual Activities Due to Asthma
Description: Defined as days not able to work or go to school because of asthma symptoms OR days not able to carry out usual activities due to asthma
Time Frame: Monthly through study completion an average of 15 months
Measure: Mean (95% Confidence Interval); unit: days per year
Arm/Group | PARTICS | Usual Care
Number analyzed (Participants) | 600 | 601
days per year | 13.4 [11.9 to 15.2] | 16.8 [14.9 to 18.9]
Statistical Analysis 1: Comparison: PARTICS vs Usual Care; Test type: Superiority — Negative binomial regression model is used, with time as an offset to account for differential duration of follow-up. The model adjusts for all the baseline covariates included in the primary analysis; Rate ratio = 0.80, 95% CI 2-sided [0.67 to 0.95]

ADVERSE EVENTS:
Time Frame: From enrollment to study completion, an average of 15 months per participant.
Description: SAE was defined as any event that resulted in death, hospitalization, persistent/significant disability, or congenital anomaly/birth defect; or was otherwise life-threatening. Data on adverse events that resulted in hospitalization or death were obtained by participant report or site report. Adverse events were not monitored/assessed with regard to the specific Adverse Event Term.
Arm/Group | PARTICS | Usual Care
All-Cause Mortality (participants affected / at risk) | 3/609 | 4/611
Serious Adverse Events (participants affected / at risk) | 75/609 | 74/611
Other Adverse Events (participants affected / at risk) | 0/609 | 0/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PARTICS (N=609) | Usual Care (N=611)
Asthma (Respiratory, thoracic and mediastinal disorders) | 43 (68) | 45 (85)
Cardiac events (Cardiac disorders) | 8 (9) | 10 (10)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (6) | 4 (4)
Hematology/oncology (Blood and lymphatic system disorders) | 0 (0) | 4 (11)
Immune system disorders (Immune system disorders) | 1 (1) | 2 (2)
Infections and infestations (Infections and infestations) | 12 (12) | 8 (9)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Nervous system disorders (Nervous system disorders) | 3 (4) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 2 (6)
Renal/urinary disorders (Renal and urinary disorders) | 2 (2) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory, thoracic, mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 2 (2) | 1 (1)
Unclassified elsewhere (General disorders) | 10 (11) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT02995733/Prot_SAP_002.pdf